CLINICAL TRIAL: NCT03118791
Title: Investigation on Acute Dose-Dependent Effects of Anthocyanins on Endothelial Function
Brief Title: Dose-Dependent Effects of Anthocyanins on Endothelial Function in Healthy Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Principal Investigator, Heinrich-Heine University, Duesseldorf
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACND
Record Dates: First submitted 2017-04-07; First posted 2017-04-18 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Healthy Men
MeSH Terms: interventions — Anthocyanins

STUDY DESIGN:
Intervention Model Description: Double blind randomized controlled crossover
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator): Capsules containing maltodextrin
  Interventions: Dietary Supplement: anthocyanins
- 80 mg ACN (Active Comparator): Capsules containing 80 mg anthocyanins
  Interventions: Dietary Supplement: anthocyanins
- 160 mg ACN (Active Comparator): Capsules containing 160 mg anthocyanins
  Interventions: Dietary Supplement: anthocyanins
- 240 mg ACN (Active Comparator): Capsules containing 240 mg anthocyanins
  Interventions: Dietary Supplement: anthocyanins
- 320 mg ACN (Active Comparator): Capsules containing 320 mg anthocyanins
  Interventions: Dietary Supplement: anthocyanins
- 480 mg ACN (Active Comparator): Capsules containing 480 mg anthocyanins
  Interventions: Dietary Supplement: anthocyanins

INTERVENTIONS:
Dietary Supplement: anthocyanins — Acute intake of capsules

SUMMARY:
Anthocyanins are a subclass of (poly)phenols very abundant in berries and red grapes. Increasing evidence from human epidemiological and dietary intervention studies suggests that anthocyanins may have cardiovascular health benefits. The present study aimes to investigate whether pure anthocyanin consumption improves endothelial function in healthy individuals and if these effects are dose-dependent.

DETAILED DESCRIPTION:
Anthocyanins are a subclass of (poly)phenols very abundant in berries and red grapes. Increasing evidence from human epidemiological and dietary intervention studies suggests that anthocyanins may have cardiovascular health benefits. A double blind randomized controlled crossover, dose-response study will be conducted in 10 young healthy men. On 6 different days, subjects will consume capsules containing 0, 80, 160, 240, 320 and 480 mg of purified anthocyanins with a one-week wash-out period. Flow-mediated dilation (FMD) and blood pressure will be measured at baseline and at 2 and 6 h after consumption. Blood samples will also be taken and quantification of plasma anthocyanin metabolites using UPLC-Q-TOF-MS will be performed. The aim is to investigate whether purified anthocyanins are able to increase FMD at 2h and 6h post consumption and whether these effects correlate with anthocyanin- derived phenolic acids quantified in the plasma.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men aged 18-45 years old
* Subjects are willing to maintain their normal eating/drinking habits and exercise habits to avoid changes in body weight over the duration of the study - subjects are able to understand the nature of the study
* able to give signed written informed consent
* signed written infomred consent form
* healthy male subjects (no clinical signs or symptoms of CVD.

Exclusion Criteria:

* cardiovascular disease, acute inflammation, cardiac arrhythmia, renal failure, heart failure (NYHA II-IV), diabetes mellitus, C-reactive protein > 0.5 mg/dL, malignant disease, hypotension (≤100 / 60 mm Hg)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Endothelial function | Changes from baseline to 2 hours postconsumption
  Flow-mediated dilation

SECONDARY OUTCOMES:
Blood pressure | 0 and 2 hours postconsumption
  Automatic measurements

OTHER OUTCOMES:
Other Pre-specified Outcome Measures | 0 and 2 hours postconsumption
  Plasma (poly)phenol metabolites measured by ultra-performance liquid chromatography quadrupole time of flight mass spectrometry (UPLC-Q-TOF MS)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, University Hospital Duesseldorf, Düsseldorf, Germany